CLINICAL TRIAL: NCT07042334
Title: Aim 3: Pilot Study of a Serious Game to Promote Transition Readiness Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Heart Association (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Rebecca Delaney, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB_00179379; 1K12TR004413 (NIH); 23SCEFIA1154397 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-06-04; First posted 2025-06-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Serious Games; Transition-age Youth; Transition to Adult Care; Congenital Heart Defect; Congenital Heart Disease in Adolescence; Patient Centered Care
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serious Game (Experimental): Receive serious game to build transition readiness skills
  Interventions: Behavioral: Serious game for transition readiness

INTERVENTIONS:
Behavioral: Serious game for transition readiness — The serious game is an interactive narrative fiction game in which players guide a character through a hospital setting, making choices that simulate real-life healthcare scenarios. The game is designed to improve skills such as communication with healthcare providers, understanding medical information, and managing appointments and medications. No drugs or medical devices are used in this intervention.

SUMMARY:
This study involves testing a new video game designed to support adolescents with congenital heart disease (CHD) in preparing to manage their health independently. The game aims to teach essential skills such as communicating with healthcare providers, understanding medical information, and managing appointments and medications. This small pilot study will evaluate the game's usability, acceptability, and its impact on participants' confidence and preparedness for managing their heart care. Feedback will be collected from adolescent participants, their parents, and healthcare providers, and the study will examine how the game influences communication during clinical visits.

ELIGIBILITY:
Inclusion criteria:

- Patient with congenital heart disease, their parent, and their clinician

Exclusion criteria:

-Significant visual or cognitive impairment that would impede their ability to play the game and/or complete the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of game logins | 1 month
  Metadata metrics from players interaction with the game will be collected, including the number of game logins. The higher the number the more engagement with the game.
Length of time spent on game | 1 month
  Metadata metrics from players interaction with the game will be collected, including the amount of time spent (i.e., minutes) on the game. The greater the amount of time the more engagement with the game.
Game sections completed | 1 month
  Metadata metrics from players interaction with the game will be collected including the number of game sections that are completed. The higher the number indicates more engagement with the game.
Recruitment of participants in the study | 1-month
  A percentage will be calculated from the number of participants approached and number of participants who enrolled to report on recruitment. Sufficient recruitment is equal to or greater than 60%.
Retention of participants | 1.5 month
  Retention of participants will be assessed by calculating a percentage from the number who enrolled and number who completed the study. Sufficient retention will be greater than or equal to 60%.
Acceptability | 1-month
  After completing the intervention, participants will be asked to complete questionnaires about their satisfaction and usability of the game (e.g., system usability scale (SUS). On the SUS, responses are from 1 to 5 for each item and greater scores indicate higher acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Children's Hospital and University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided